CLINICAL TRIAL: NCT05575713
Title: The Predictive Effect of Soluble Epoxide Hydrolase (SEH) on Depression Treatment, Cognition and Suicide Improvement
Brief Title: The Effect of Soluble Epoxide Hydrolase (SEH) on Depression
Status: Completed | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2022-092
Record Dates: First submitted 2022-08-28; First posted 2022-10-12 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Major Depressive Disorder
Keywords: depression; cognition; suicide; Soluble epoxide hydrolase，sEH; prediction
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Suicide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Major depressive disorder: Patients diagnosed with severe depressive episode according to the diagnostic and Statistical Manual of mental disorders, 5th Edition (DSM-V);
- healthy volunteer: Person who did not meet the DSM-V diagnosis of any mental disease, had no family history of psychiatric disease, and had no history of suicidal behavior.

SUMMARY:
Depression is the most common mental disease and the second leading cause of chronic disease burden, which is closely related to suicidal behavior. The diagnosis and treatment of depression still lack of effective biological indicators, and about 30% of patients with depression still can not relieve their depressive symptoms after treatment. Previous studies have found that ATP release from astrocytes plays an important role in the occurrence, development and treatment of depression. Epoxy eicosotrienes (eets) are closely related to the function of the nervous system and may be the pathophysiological mechanism of depression. Soluble epoxide hydrolase (SEH) can regulate ATP release by affecting EET degradation, leading to depression like behavior and antidepressant effect, and sEH is closely related to cognitive function of depression.

DETAILED DESCRIPTION:
This study is an observational study without any intervention treatment for the subjects. All subjects need to sign the informed consent before screening, and the successful subjects can enter the study. Routine clinical diagnosis and treatment were performed on patients with depression, and the treatment effect of depressive symptoms, neurocognitive function and suicide improvement were evaluated at the 2nd week, 1st, 2nd, 3rd, 6th and 12th months after enrollment, and statistical analysis was conducted. The treatment lasted until the subjects completed the 12th month follow-up or reached any of the withdrawal criteria. This study will clarify the relationship between sEH gene polymorphism and mRNA expression and depression and suicide behavior, and explore the predictive role of soluble epoxide hydrolase sEH in the treatment effect of depression, cognition and suicide improvement during the follow-up study.

ELIGIBILITY:
* Inclusion criteria:

  1. Voluntarily sign informed consent;
  2. Age: 18-65 years old;
  3. Elementary school or above, able to understand and complete all inspections and assessments;
  4. Did not take any psychotropic drugs (including benzodiazepines) within 2 weeks before enrollment;
  5. After routine medical diagnosis by clinicians, they were divided into depression and healthy people.
* Exclusion criteria:

  1. Severe somatic or neurological diseases;
  2. Mental retardation and dementia;
  3. During pregnancy or breastfeeding;
  4. Heavy smoking, alcoholism and other substance abuse or dependence (within 3 months before enrollment);
  5. Electric shock treatment (within 3 months before enrollment);
  6. According to the judgment of the investigator, it is not suitable to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with major depressive disorder in the outpatient department of psychiatry and psychology of Nanfang Hospital
Sampling Method: Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Hamilton Depression Scale (HAMD-24) | Baseline, the second week, the first month, the second month, the third month, the sixth month and the first year
  Scores ranging from 0-76, with higher scores indicate more severe symptoms

SECONDARY OUTCOMES:
Change in Columbia-Suicide Severity Rating Scale, C-SSRS | Baseline, the second week, the first month, the second month, the third month, the sixth month and the first year
  Scores ranging from 0-42, with higher scores indicate more severe symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Honglei Yin, doctor, Study Chair — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zheng S, Guo J, Zheng R, Ji Y, Zhong Q, Yin H. A Naturalistic Prospective Study of the Prognostic Impact of EPHX2 in Major Depressive Disorder: Impulsivity may be an Important Factor. Depress Anxiety. 2025 Apr 13;2025:8124403. doi: 10.1155/da/8124403. eCollection 2025. PMID 40259894
- [Derived] Zheng S, Zeng W, Wu Q, Li W, He Z, Li E, Tang C, Xue X, Qin G, Zhang B, Yin H. Predictive Models for Suicide Attempts in Major Depressive Disorder and the Contribution of EPHX2: A Pilot Integrative Machine Learning Study. Depress Anxiety. 2024 May 9;2024:5538257. doi: 10.1155/2024/5538257. eCollection 2024. PMID 40226652
- [Derived] Ji Y, Liu X, Zheng S, Zhong Q, Zheng R, Huang J, Yin H. Validation and application of the Chinese version of the Columbia-Suicide Severity Rating Scale: Suicidality and cognitive deficits in patients with major depressive disorder. J Affect Disord. 2023 Dec 1;342:139-147. doi: 10.1016/j.jad.2023.09.014. Epub 2023 Sep 14. PMID 37714386

DOCUMENTS (1):
  • Study Protocol (2022-05-25): https://cdn.clinicaltrials.gov/large-docs/13/NCT05575713/Prot_000.pdf